CLINICAL TRIAL: NCT02321969
Title: Green Tea Extracts for the Prevention of Colorectal Adenomas and Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B-1006/103-002
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Neoplasms, Colorectal
Keywords: Chemoprevention; Colorectal adenomatous polyp; Green tea extract
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Without green tea extract (GTE) supplementation
- GTE group (Experimental): GTE supplementation for 12 months after polypectomy for colorectal adenomatous polyps
  Interventions: Dietary Supplement: GTE (green tea extract)

INTERVENTIONS:
Dietary Supplement: GTE (green tea extract) — 6 GTE tablets per day. Daily dose is equivalent of 9 cup-of-green tea per day (0.9 g/day GTE, 0.6 g/day epigallocatechin gallate [EGCG]).
  Arms: GTE group

SUMMARY:
Experimental studies have shown the chemopreventive properties of green tea extract (GTE) on colorectal cancer. And colorectal adenomas are precursors to colorectal cancers. The aim of this study is to determine the preventive effect of GTE supplements on metachronous colorectal adenomas by giving GTE tablets of which are equivalent of 9 cup-of-green tea per day (0.9 g/day GTE, 0.6 g/day Epigallocatechin gallate (EGCG).

DETAILED DESCRIPTION:
The subjects who had undergone complete removal of colorectal adenomas by endoscopic polypectomy have been enrolled since June 2010. They were then randomized into two groups as follows: supplementation group (0.9 g GTE per day for 12 months) or control group without GTE supplementation. Follow-up colonoscopy was conducted in 12 months. A structured 72-h recall at baseline and the 1-year follow-up was used to assess dietary factors, and to evaluate rectal mucosal proliferation index (RMPI) using known proliferation markers (Ki-67/PCNA), at least 2 random biopsies of rectal mucosa were taken. A sample size of 176 patients (88 per each group) was calculated to give the study 80% power to detect a difference, assuming a two-sided significance test at the 0.05 level.

ELIGIBILITY:
Inclusion Criteria:

- subjects who present one or more adenomatous polyps on colonoscopy.

Exclusion Criteria:

* subjects who denied to participate in this study
* subjects who present inflammatory bowel diseases such as ulcerative colitis or crohn's disease
* subjects who received partial or total colectomy due to colon cancer or other colonic diseases.
* subjects who are pregnant
* subjects who are on aspirin or NSAIDS for any reasons
* subjects who have received a transplant of any major organ or who are on immunosuppressants for any reason
* subjects who are unable to perform a bowel prep or who present poor bowel prep for colonoscopy

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2010-08; Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Recurrence/Number/Size of metachronous colorectal adenoma(s) | 1 year

SECONDARY OUTCOMES:
Recurrence/Number/Size of metachronous colorectal polyp(s) including hyperplastic polyp(s) | 1 year
Change of lipid profiles after green tea extract (GTE) supplementation | 1 year
Change of body weight, BMI and waist circumference | 1 year
Adverse effect(s) of GTE supplementation | every 1-3 months till the end of study protocol (12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Dong Ho Lee, M.D., Ph.D., Principal Investigator — Seoul National Universtiy Bundang Hospital

REFERENCES:
- [Result] Shimizu M, Fukutomi Y, Ninomiya M, Nagura K, Kato T, Araki H, Suganuma M, Fujiki H, Moriwaki H. Green tea extracts for the prevention of metachronous colorectal adenomas: a pilot study. Cancer Epidemiol Biomarkers Prev. 2008 Nov;17(11):3020-5. doi: 10.1158/1055-9965.EPI-08-0528. PMID 18990744
- [Result] Stingl JC, Ettrich T, Muche R, Wiedom M, Brockmoller J, Seeringer A, Seufferlein T. Protocol for minimizing the risk of metachronous adenomas of the colorectum with green tea extract (MIRACLE): a randomised controlled trial of green tea extract versus placebo for nutriprevention of metachronous colon adenomas in the elderly population. BMC Cancer. 2011 Aug 18;11:360. doi: 10.1186/1471-2407-11-360. PMID 21851602
- [Derived] Shin CM, Lee DH, Seo AY, Lee HJ, Kim SB, Son WC, Kim YK, Lee SJ, Park SH, Kim N, Park YS, Yoon H. Green tea extracts for the prevention of metachronous colorectal polyps among patients who underwent endoscopic removal of colorectal adenomas: A randomized clinical trial. Clin Nutr. 2018 Apr;37(2):452-458. doi: 10.1016/j.clnu.2017.01.014. Epub 2017 Jan 29. PMID 28209333